CLINICAL TRIAL: NCT02814929
Title: Incidence, Risk Factors and Severity of Retinopathy of Prematurity (ROP) in Turkey: A Prospective Multicenter Study Including 69 NICUs
Brief Title: Incidence, Risk Factors and Severity of Retinopathy of Prematurity (ROP) in Turkey
Acronym: TR-ROP
Status: Completed | Type: Observational
Sponsor: Etlik Zubeyde Hanım Women's Health Care, Training and Research Hospital (Other)
Collaborators: Acibadem Atakent University Hospital (Other); Baskent University (Other); Adana Numune Training and Research Hospital (Other Government); Aydin Adnan Menderes University (Other); Ankara University (Other); Baskent University Ankara Hospital (Other); Ankara Guven Hospital (Unknown); Ataşehir Kadıkoy Sifa Hospital (Unknown); Ataturk University (Other); Bagcilar Training and Research Hospital (Other Government); Bezmialem Vakif University (Other); Dortcelik Children Hospital (Unknown); Uludag University (Other); Bulent Ecevit University (Other); Canakkale 18 Mart University (Unknown); Cukurova University (Other); Denizli Devlet Hastanesi (Other); Denizli Ozel Saglik Hospital (Unknown); Dicle University (Other); Dokuz Eylul University (Other); Doruk Bursa Hospital (Unknown); Faruk Sukan Maternity and Children Hospital (Unknown); Ege University (Other); Erzurum Nenehatun Maternity Hospital (Unknown); Eskisehir Osmangazi University (Other); Firat University (Other); Cengiz Gokcek Women's and Children's Hospital (Other); University of Gaziantep (Other); Mustafa Kemal University (Other); Hacettepe University (Other); Istanbul Medeniyet University (Other); Istanbul Medipol University Hospital (Other); Istanbul University (Other); Dr. Behcet Uz Children's Hospital (Other); Kahramanmaras Megapark Hospital (Other); Kahramanmaras Sutcu Imam University (Other); Kanuni Sultan Suleyman Training and Research Hospital (Other); Karadeniz Technical University (Other); TC Erciyes University (Other); Kecioren Education and Training Hospital (Other); Kırıkkale University (Other); Konya Baskent University (Unknown); Konya Meram State Hospital (Other); Selcuk University (Other); Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government); Marmara University (Other); Medical Park Gaziantep Hospital (Other); Mersin Maternity Hospital (Unknown); NCR International Hospital (Unknown); Necmettin Erbakan University (Other); Ozel Medova Hospital (Unknown); Pamukkale University (Other); Umraniye Education and Research Hospital (Other Government); Inonu University (Other); Sami Ulus Maternity and Children Hospital (Unknown); Ondokuz Mayıs University (Other); Suleymaniye Birth And Women's Health Education And Research Hospital (Other Government); Sisli Hamidiye Etfal Training and Research Hospital (Other); Tepecik Training and Research Hospital (Other); Tokat Gaziosmanpasa University (Other); Trabzon Kanuni Education and Research Hospital (Other); Trakya University (Other); Yuksek Ihtisas University (Other); Yuzuncu Yil University (Other); Zekai Tahir Burak Women's Health Research and Education Hospital (Other); Zeynep Kamil Maternity and Pediatric Research and Training Hospital (Other); Muğla Sıtkı Koçman University (Other); Koç University (Other)
Responsible Party: Principal Investigator, Ahmet Yagmur BAS, Neonatologist, Ankara Yildirim Beyazıt University
Other Study IDs: Turkey ROP Study
Record Dates: First submitted 2016-06-14; First posted 2016-06-28 (Estimated); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Retinopathy of Prematurity
Keywords: ROP; Risk factors; Incidence; Turkey
MeSH Terms: conditions — Retinopathy of Prematurity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Demographic and Prenatal Characteristics: Gender, multiple pregnancy antenatal steroid therapy, invitro fertilisation, preeclampsia/eclampsia, infants of diabetic mother, chorioamnionitis will be compared among infants with and without ROP
- Neonatal Characteristics of infants: Neonatal characteristics: GA, BW, SGA, resuscitation in delivery room, RDS, duration of mechanical ventilation and oxygen therapy, intracranial hemorrhage, hemodynamically significant PDA, early/late sepsis, NEC, number of blood transfusions, BPD, breastfeeding and weight gain at postnatal 28th day will be compared among infants with and without ROP.
- Incidence of any ROP and severe ROP: Incidence of any ROP, severe ROP and its treatment in relation to BW and GA will be evaluated. The same parameters will also be evaluated in preterm babies of refugees.

SUMMARY:
The study includes preterm infants who are being screened for ROP between April 1,2016 and April 30, 2017 in 69 neonatal intensive care units (NICUs) in Turkey. Infants with birth weight (BW) of ≤1500 g or ≤32 weeks' gestation and those with a BW of greater than 1500 g or gestational age (GA) >32 weeks with an unstable clinical course are included. The incidence of any ROP, severe ROP and treatment modalities will be determined. The risk factors for ROP development will also be evaluated.

DETAILED DESCRIPTION:
This study, promoted by the "Turkish Neonatology Society", involved preterm infants who are being screened for ROP between April 1, 2016 and April 30, 2017 in level III Turkish NICUs.

An electronic questionnaire is being filled by certified neonatologists in Turkey via a special network. Neonatologists working in 69 centers who agreed to participate in this study provide their data regarding the ROP in their NICU. The medical records of retinal examinations of preterm infants who met the screening criteria will be evaluated.

A case report form for each patient will be filled including risk factors for the development of ROP such as gestational age, birth weight, small for gestational age (SGA), gender, multiple gestation, antenatal steroid therapy, invitro fertilisation, preeclampsia/eclampsia, infants of diabetic mother, chorioamnionitis, resuscitation in delivery room, respiratory distress syndrome (RDS), duration of mechanical ventilation and oxygen therapy, intracranial hemorrhage, hemodynamically significant patent ductus arteriosus (PDA), early/late sepsis, necrotising enterocolitis (NEC), number of blood transfusions, bronchopulmonary dysplasia (BPD), weight gain at postnatal 28th days and breastfeeding.

Risk factors for developing ROP will be evaluated. Multivariate analysis will be performed among significant variables.

In addition, the incidence of any ROP, severe ROP in relation to GA and BW and treatment modalities will be determined. Severe ROP is defined as ROP requiring treatment.

Since Turkey is receiving many refugees in recent years, the investigators also planned to evaluate the incidence and risk factors for developing ROP in preterm babies of refugees.

Ophthalmologic examination is continued until full vascularisation. So, the maximum stage of ROP detected for every infant will be reported. Data from 69 NICUs will be pooled together and analyzed.

The "International Classification of ROP" guidelines are used to record stage of disease, location by zone, signs of plus disease and signs of regression. Criteria for treatment of ROP are based on the Early Treatment for Retinopathy of Prematurity (ETROP) recommendation. Confirmed forms are also assigned by the parents before the initial screening and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Infants with BW ≤1500 g or ≤32 weeks' gestation and those with a BW of greater than 1500 g or GA >32 weeks requiring cardiorespiratory support and who were determined by the attending clinician to be at risk for ROP, are included.

Exclusion Criteria:

* Neonates who died before the first ROP examination are excluded from the study.

Min Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Preterm babies screened for ROP.
Sampling Method: Non-Probability Sample
Enrollment: 6115 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-10-17 (Actual)

PRIMARY OUTCOMES:
Incidence of ROP in Turkey | 12 months
  Incidence of ROP and severe ROP in relation to GA and BW in Turkey

SECONDARY OUTCOMES:
The association of antenatal corticosteroid administration with ROP | 12 months
The role of sepsis in infants in the development of ROP | 12 months
  Culture proven and clinical early and late sepsis will be evaluated
The relationship between rate of postnatal weight gain and severity of ROP | 12 months
The relationship between breastfeeding and ROP development | 12 months
ROP in SGA premature infants | 12 months
  Comparison of ROP in SGA infants with those of appropriate size for GA
ROP in multiple births | 12 months
  Comparison of the frequency and severity of ROP among singleton and multiple-birth neonates
The role of transfusions in ROP development | 12 months
Duration of oxygen therapy among infants with and without ROP | 12 months
Number of patients requiring laser photocoagulation treatment | 12 months
Number of patients requiring vitreoretinal surgery | 12 months
Number of patients requiring anti-vascular endothelial growth factor treatment | 12 months

OTHER OUTCOMES:
Incidence of ROP in preterm babies of refugees in Turkey | 12 months
  Incidence of any ROP and severe ROP in relation to GA and BW in preterm babies of refugees

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Y Bas, MD, Principal Investigator — Etlik Zubeyde Hanim Womens' Health and Teaching Hospital; Nihal Demirel, MD, Principal Investigator — Etlik Zubeyde Hanim Womens' Health and Teaching Hospital; İbrahim M Hirfanoglu, MD, Principal Investigator — Gazi University; Dilek U Isik, MD, Principal Investigator — Etlik Zubeyde Hanim Womens' Health and Teaching Hospital; Turan Tunc, MD, Principal Investigator — Istanbul; Esin Koc, MD, Principal Investigator — Gazi University
Locations (1):
- Etlik Zubeyde Hanim Womens' Health and Teaching Hospital, Ankara, Keçi̇ören, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bas AY, Koc E, Dilmen U; ROP Neonatal Study Group. Incidence and severity of retinopathy of prematurity in Turkey. Br J Ophthalmol. 2015 Oct;99(10):1311-4. doi: 10.1136/bjophthalmol-2014-306286. Epub 2015 Apr 13. PMID 25868788
- [Derived] Bas AY, Demirel N, Koc E, Ulubas Isik D, Hirfanoglu IM, Tunc T; TR-ROP Study Group. Incidence, risk factors and severity of retinopathy of prematurity in Turkey (TR-ROP study): a prospective, multicentre study in 69 neonatal intensive care units. Br J Ophthalmol. 2018 Dec;102(12):1711-1716. doi: 10.1136/bjophthalmol-2017-311789. Epub 2018 Mar 8. PMID 29519879